CLINICAL TRIAL: NCT03258333
Title: Small Aortic Annulus - a New Solution to the Old Problem
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The Federal Centre of Cardiovascular Surgery, Russia (Other)
Responsible Party: Principal Investigator, Mikulyak Artur, Principal Investigator, Cardiovascular surgeon, The Federal Centre of Cardiovascular Surgery, Russia
Other Study IDs: FederalCCS002
Record Dates: First submitted 2017-07-23; First posted 2017-08-23 (Actual); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Aortic Valve Replacement
Keywords: aortic stenosis, aortic valve replacement, pericardium
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stented bioprosthesis: Standard aortic valve replacement with stented bioprosthesis. Surgery is performed through median sternotomy, aortic and right or bicaval venous cannulation, normothermic perfusion, antegrade cardioplegia with use cardioplegic solution Custodiol. A transverse aortotomy was performed 1 to 2 cm above the right coronary artery. The aortic annulus was thoroughly débrided of calcium. Valve sizing was performed with standard manufacturers' sizers, with selection of the size that would comfortably fit within the aortic annulus. A noneverting suture technique was used in all patients with interrupted horizontal mattress 2-0 braided sutures placed around the aortic annulus, with the pledgets on the ventricular aspect.
  Interventions: Procedure: aortic valve replacement
- Ozaki procedure: Aortic valve reconstruction using autologus pericardium (Ozaki procedure). The autologous pericardium is harvested after routine median sternotomy. Harvested pericardium is then treated with a 0.6% glutaraldehyde solution for 10 min and then rinsed 3 times with sterilized saline each time for 6 min. After resection of the diseased aortic valve cusps, the distance between each commissure is measured using a self-developed sizing instrument. Glutaraldehyde-treated autologous pericardium is trimmed with a self-developed template corresponding to the measured value. The annular margin of the pericardial leaflet is then running-sutured to each annulus with 3-0 monofilament sutures. Commissural coaptation is secured with additional 4-0 monofilament sutures. The coaptation of the 3 cusps is then checked with negative pressure on the left ventricular vent.
  Interventions: Procedure: aortic valve replacement

INTERVENTIONS:
Procedure: aortic valve replacement — Standart AVR using stented stented bioprosthesis aortic valve reconstruction using autologus pericardium

SUMMARY:
In this prospective single-center study included 60 patients with a severe degenerative aortic stenosis and small aortic annulus (<21 mm) who underwent standard AVR with stented bioprosthesis (group 1, n=30) and aortic valve reconstruction using autologus pericardium (Ozaki procedure) (group 2, n=30)

DETAILED DESCRIPTION:
Aortic valve replacement (AVR) in patients with a small aortic annulus is a challenging problem. Implantation of a small aortic valve sometimes leads to high residual gradients, despite a normally functioning prosthesis. Patients with a small aortic annulus, especially those with a large body surface area, are at higher risk of prosthesis-patient mismatch, which is associated with worse clinical outcomes and decreased survival. The purpose of this study was to compare the hemodynamic performance among the 2 management strategies (standard AVR with stented bioprosthesis and Ozaki procedure) in the context of a small aortic annulus (<21 mm)

ELIGIBILITY:
Inclusion Criteria:

* severe degenerative aortic valve stenosis

Exclusion Criteria:

* redo operation, infective endocarditis

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe degenerative aortic stenosis and small aortic annulus (<21 mm) were enrolled in this study
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-02-18 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Indexed effective orifice area, cm²/m² | 12 months after surgery
  Assessment of aortic valve dimension

SECONDARY OUTCOMES:
prosthesis-patient mismatch (PPM) | 12 months after surgery
  Indicator of the effectiveness of aortic valve replacement
Peak pressure gradient, mm.Hg | 12 months after surgery
  Indicator of the effectiveness of aortic valve replacement
Mean pressure gradient, mm.Hg | 12 months after surgery
  Indicator of the effectiveness of aortic valve replacement
Effective orifice area, EOA, cm² | 12 months after surgery
  Assessment of aortic valve dimension

OTHER OUTCOMES:
Age (years) | 12 months after surgery
  Description and comparison of groups patients
Body mass index, kg/m² | 12 months after surgery
  Description and comparison of groups patients
Body surface area, m² | 12 months after surgery
  Description and comparison of groups patients
Aortic annulus diameter, mm | 12 months after surgery
  Description and comparison of groups patients
Indexed aortic annulus diameter, mm/m² | 12 months after surgery
  Description and comparison of groups patients
Myocardial mass index, g/m² | 12 months after surgery
  Assessment of reverse remodeling of the left ventricle

CONTACTS AND LOCATIONS:
Locations (1):
- FederalCCS, Penza, Russia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Gerosa G, Tarzia V, Rizzoli G, Bottio T. Small aortic annulus: the hydrodynamic performances of 5 commercially available tissue valves. J Thorac Cardiovasc Surg. 2006 May;131(5):1058-64. doi: 10.1016/j.jtcvs.2005.12.034. PMID 16678590
- [Result] Ozaki S, Kawase I, Yamashita H, Uchida S, Takatoh M, Hagiwara S, Kiyohara N. Aortic Valve Reconstruction Using Autologous Pericardium for Aortic Stenosis. Circ J. 2015;79(7):1504-10. doi: 10.1253/circj.CJ-14-1092. Epub 2015 Mar 30. PMID 25818901
- [Result] Ozaki S, Kawase I, Yamashita H, Uchida S, Nozawa Y, Matsuyama T, Takatoh M, Hagiwara S. Aortic valve reconstruction using self-developed aortic valve plasty system in aortic valve disease. Interact Cardiovasc Thorac Surg. 2011 Apr;12(4):550-3. doi: 10.1510/icvts.2010.253682. Epub 2011 Jan 27. PMID 21273254
- [Result] Borger MA, Nette AF, Maganti M, Feindel CM. Carpentier-Edwards Perimount Magna valve versus Medtronic Hancock II: a matched hemodynamic comparison. Ann Thorac Surg. 2007 Jun;83(6):2054-8. doi: 10.1016/j.athoracsur.2007.02.062. PMID 17532395
- [Result] Ghoneim A, Bouhout I, Demers P, Mazine A, Francispillai M, El-Hamamsy I, Carrier M, Lamarche Y, Bouchard D. Management of small aortic annulus in the era of sutureless valves: A comparative study among different biological options. J Thorac Cardiovasc Surg. 2016 Oct;152(4):1019-28. doi: 10.1016/j.jtcvs.2016.06.058. Epub 2016 Jul 28. PMID 27641297
- [Result] Morita S. Aortic valve replacement and prosthesis-patient mismatch in the era of trans-catheter aortic valve implantation. Gen Thorac Cardiovasc Surg. 2016 Aug;64(8):435-40. doi: 10.1007/s11748-016-0657-9. Epub 2016 May 27. PMID 27234223
- [Result] Minardi G, Pergolini A, Zampi G, Pulignano G, Pero G, Sbaraglia F, Pino PG, Cioffi G, Musumeci F. St. Jude Trifecta versus Carpentier-Edwards Perimount Magna valves for the treatment of aortic stenosis: comparison of early Doppler-echocardiography and hemodynamic performance. Monaldi Arch Chest Dis. 2013 Sep;80(3):126-32. doi: 10.4081/monaldi.2013.74. PMID 24818319